CLINICAL TRIAL: NCT01040351
Title: Effect of Ultrasound Guided Aspiration of Hydrosalpingeal Fluid at the Time of Oocyte Retrieval on the Outcomes of IVF-ET, a Randomized Controlled Trial
Brief Title: Ultrasound Guided Aspiration of Hydrosalpingeal Fluid and IVF-ET Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Ahmed Elgazzar Hospital (Other)
Responsible Party: Usama Fouda , MD, PhD, Cairo university.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hydrosalpinx1
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2010-10

CONDITIONS: Infertility
Keywords: Infertility; Hydrosalpinx; IVF-ET
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Hydrosalpinx needle aspiration (Experimental): After the retrieval of oocytes an aspiration needle is inserted into the hydrosalpinx under ultrasonographic guidance and suction is applied to aspirate the hydrosalpingeal fluid completely .
  Interventions: Procedure: ultrasound guided aspiration of hydrosalpingeal fluid
- 2. no aspiration (No Intervention): IVF-ET is done without prior aspiration of hydrosalpingeal fluid

INTERVENTIONS:
Procedure: ultrasound guided aspiration of hydrosalpingeal fluid — Under deep sedation, the retrieval of oocytes is done and then an aspiration needle is inserted into the hydrosalpinx under ultrasonographic guidance and suction is applied to aspirate the hydrosalpingeal fluid completely . If there are bilateral hydrosalpinges, the process is repeated on the opposite side.
  Other Names: ultrasound guided Hydrosalpinx needle aspiration
  Arms: 1: Hydrosalpinx needle aspiration

SUMMARY:
The aim of this study is to determine whether the ultrasound guided aspiration of hydrosalpingeal fluid at the time of oocyte retrieval can improve the outcomes of IVF-ET .

DETAILED DESCRIPTION:
A Cochrane review of prospective randomized trials of laparoscopic salpingectomy confirmed the beneficial effect of laparoscopic salpingectomy on IVF ET outcomes in patients with hydrosalpinges. Surgery is not usually safe especially in patients with extensive adhesions, morbid obesity and previous multiple laparotomies. Other less invasive options for patients with hydrosalpinges as ultrasound guided aspiration of hydrosalpingeal fluid, antibiotics and hysteroscopic occlusion of fallopian tube were studied in order to find an alternative to salpingectomy. Although these methods are simple and getting popular,current data are inadequate to recommend these treatment options instead of salpingectomy. The aim of this study is to determine whether the ultrasound guided aspiration of hydrosalpingeal fluid at the time of oocyte retrieval can improve the outcomes of IVF-ET .

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral hydrosalpinges visible by ultrasound
* Age between 18 - 37 years
* Period of infertility > 1 year
* Body mass index between 19-29
* Normal basal luteinizing hormone (LH), follicle stimulating hormone (FSH) and prolactin concentrations
* Normal recent semen analysis (according to World Health Organization criteria)

Exclusion Criteria:

* Uterine fibroid requiring surgical removal
* Endometriosis
* Male factor of infertility requiring ICSI
* Previous IVF cycles
* History of recurrent miscarriage
* Endocrinologic disorders
* Presence of systemic disease contraindicating pregnancy

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2006-10; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D, PhD, Study Chair — Lecturer of obstetrics and Gynecology , Faculty of medicine ,Cairo university.; Ahmed M sayed, MD,PhD, Study Director — Assistant professor of obstetrics and Gynecology , Faculty of medicine ,Cairo university.
Locations (1):
- Ahmed Elgazzar hospital , Assisted conception unit, Giza, 35 Eleshreen Saint King Faisal., Egypt

REFERENCES:
- [Background] Hammadieh N, Coomarasamy A, Ola B, Papaioannou S, Afnan M, Sharif K. Ultrasound-guided hydrosalpinx aspiration during oocyte collection improves pregnancy outcome in IVF: a randomized controlled trial. Hum Reprod. 2008 May;23(5):1113-7. doi: 10.1093/humrep/den071. Epub 2008 Mar 13. PMID 18343810
- [Derived] Fouda UM, Sayed AM. Effect of ultrasound-guided aspiration of hydrosalpingeal fluid during oocyte retrieval on the outcomes of in vitro fertilisation-embryo transfer: a randomised controlled trial (NCT01040351). Gynecol Endocrinol. 2011 Aug;27(8):562-7. doi: 10.3109/09513590.2010.507290. Epub 2010 Jul 30. PMID 20672903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was two arm prospective randomized controlled study including 110 fresh IVF- ETs from 110 patients , undertaken between October 2006 to May 2010 at the assisted conception unit of Ahmed Elgazzar hospital , Cairo , Egypt.
Period: Overall Study
Arm/Group | 1: Hydrosalpinx Needle Aspiration | 2. no Aspiration
Started | 55 (October 2006) | 55 (October 2006)
Completed | 54 (May 2010) | 53 (May 2010)
Not Completed | 1 | 2
Not completed — poor ovarian response | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Hydrosalpinx Needle Aspiration | 2. no Aspiration | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 55 | 110
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.16 (3.6) | 29.38 (4.0) | 28.77 (3.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Achieved Clinical Pregnancy in a Transfer Cycle
Description: The Number of Participants Who Achieved Clinical Pregnancy( presence of intrauterine gestational sac detected by transvaginal ultrasound
  )in a transfer cycle
Time Frame: 5 weeks after embryo transfer
Population: Patients undergoing embryo transfer were included in final analysis
Measure: Number; unit: participents
Arm/Group | 1: Hydrosalpinx Needle Aspiration | 2. no Aspiration
Number analyzed (Participants) | 54 | 53
participents | 17 | 7
Statistical Analysis 1: Comparison: 1: Hydrosalpinx Needle Aspiration vs 2. no Aspiration; Test type: Non-Inferiority or Equivalence — . The aggregate result of 6 studies reporting the pregnancy rate of patients with ultrasound visible hydrosalpinx revealed that clinical pregnancy rate among the patients with ultrasound-visible hydrosalpinges was 12.6%. We assumed that the aspiration of hydrosalpinx could restore clinical pregnancy rate to that expected for patients with tubal factor of infertility but without hydrosalpinges (about 36.5% in our hospital); p = 0.023, Chi-squared; Odds Ratio (OR) = 3.02, 95% CI 2-sided [1.13 to 8.0]

2. Secondary Outcome: The Number of Participants Who Achieved Ongoing Pregnancy in a Transfer Cycle .
Description: The number of participants who Achieved Ongoing pregnancy (pregnancy for more than 18 weeks after embryo transfer) in a transfer cycle .
Time Frame: 18 weeks after embryo transfer
Population: Patients who underwent embryo transfer were included in the final analysis
Measure: Number; unit: participents
Arm/Group | 1: Hydrosalpinx Needle Aspiration | 2. no Aspiration
Number analyzed (Participants) | 54 | 53
participents | 15 | 5

ADVERSE EVENTS:
Time Frame: October 2006 to May 2010
Groups:
- 1: Hydrosalpinx Needle Aspiration: Aspiration of hydrosalpingeal fluid prior to IVF-ET
- 2. no Aspiration: IVF-ET without any prior intervention
Arm/Group | 1: Hydrosalpinx Needle Aspiration | 2. no Aspiration
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 0/54 | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Hydrosalpinx Needle Aspiration (N=54) | 2. no Aspiration (N=53)
Flaring of pelvic infection and peritonitis (Reproductive system and breast disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Hydrosalpinx Needle Aspiration (N=54) | 2. no Aspiration (N=53)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Several patients refused to participate in the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes